CLINICAL TRIAL: NCT05970913
Title: The Value of PET-CT in Predicting Segement Specific Lymph Nodes Metastasis in Non Small Cell Lung Cancer
Brief Title: PET-CT Predicting Segement Specific Lymph Nodes Metastasis
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Chief of the MDT board of thoracic cancer, Fudan University
Other Study IDs: ECTOP-1017
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer; Lymph Node Metastasis; Positron Emission Tomography
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter prospective clinical study that aims to evaluate the predictive value of preoperative PET-CT results (such as SUV uptake, size of tumor lymph nodes, and differences in FDG uptake compared to surrounding tissues) for lymph node metastasis in patients with non-small cell lung cancer. During surgery, all patients underwent systematic mediastinal lymph node dissection. The final pathological results were used to assess the predictive value of PET-CT for segment-specific lymph node metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Solitary tumor, or multiple tumors with only ground-glass nodules (GGNs) apart from the primary lesion.
* Diameter of the primary lesion ≤5cm, with a CTR between 0.5 and 1.
* No enlarged mediastinal lymph nodes observed on preoperative contrast-enhanced CT.
* Pathological confirmation of non-small cell lung cancer (NSCLC) either before or during surgery.
* Systematic lymph node dissection performed during surgery.
* No prior radiotherapy or chemotherapy for initial treatment.
* No history of malignant tumors.

Exclusion Criteria:

* Locally advanced or distant metastasis.
* Pleural dissemination observed during surgery.
* History of malignant tumors.
* Received neoadjuvant therapy.
* Systematic lymph node dissection not performed during surgery.
* Histopathological examination reveals lung malignancies other than non-small cell lung cancer (NSCLC).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had non small cell lung cancer received surgery and systematic lymph node dissection.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Predictive value of PET-CT for segment-specific lymph node metastasis | Preoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Shanghai, China